CLINICAL TRIAL: NCT01334099
Title: Phase I Study of Local Radiation and CP-675,206 Administration in Patients With Inoperable Locally Recurrent or Metastatic Breast Cancer
Brief Title: Safety Study of Radiation and CP-675,206 Infusion for Breast Cancer Patients
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Contract with drug supplier expired and was not renewed.
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GA3671RD IIR#1
Record Dates: First submitted 2011-01-18; First posted 2011-04-12 (Estimated); Last update posted 2015-06-22 (Estimated); Status verified 2015-06

CONDITIONS: Metastatic Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — tremelimumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Radiation combined with CP-675,206 (Experimental)
  Interventions: Biological: CP-675,206; Radiation: External local radiation therapy

INTERVENTIONS:
Biological: CP-675,206 — Intravenous infusion for one cycle (further cycles permitted as per medical assessment). Patient assigned dose of 3mg/kg, 6mg/kg, 10mg/kg, or 15mg/kg.
Radiation: External local radiation therapy — One cycle of 2000cGy administered locally to one site over 5 days.

SUMMARY:
The purpose of this study is to determine the maximum dose of CP-675,206 when given in combination with radiation. Patients will be given local radiation to one tumor site and an intravenous infusion of CP-675,206.

DETAILED DESCRIPTION:
Breast cancer is the most common cancer in Canadian women. In 2007 an estimated 22,300 women will be diagnosed and 5300 will die of the disease. Despite advances in therapy, metastatic disease remains an incurable illness, with a median survival of only 2 years. Standard systemic treatment options for metastatic disease include chemotherapy or hormonal therapy. Radiation is frequently used in the metastatic setting for palliation of symptoms, with the most frequent site of radiation being bone. Response rates to first line chemotherapy are in the range of 30%, however these responses are not durable. Currently there are no curative options for metastatic disease, underscoring the need for novel therapeutic approaches.

CTLA4 is a receptor expressed on the surface of activated T cells and regulatory T cells. CTLA-blockade has been tested in clinical trials using humanized monoclonal antibodies, and some biological responses have been reported. The anti-tumor immune response may be further augmented by the combination of CTLA4-blockade with radiation, with the potential to mediate regression of metastases outside of the field of radiation. The primary goal of this study therefore is to establish the safety of CTLA4-blockade using the antibody CP-675, 206 in combination with radiation. This trial is being conducted as a prelude to a planned phase II trial of CP-675,206 in combination with radiation in metastatic breast cancer.

ELIGIBILITY:
Inclusion Criteria:

* Inoperable locally recurrent or metastatic breast cancer
* Performance status 0-1
* Adequate organ function as determined by lab tests
* Greater than 3 weeks since any chemotherapy treatment
* Greater than 2 weeks since last dose of hormonal therapy

Exclusion Criteria:

* Previous treatment with any anti-CTLA4 agent
* Patients with active diarrhea
* Patients who will receive radiation to pelvic lesions
* History of chronic inflammatory or autoimmune disorder
* History of insulin-dependent diabetes
* History in the last 5 years of any chronic gastrointestinal conditions
* History within the last year of congestive heart failure, stroke, myocardial infarction or thromboembolic event
* Patients with known brain metastasis
* Concurrent treatment with immunosuppressive medication for longer than 10 days within 4 weeks of enrollment or while on trial
* Patients of reproductive potential not using effective contraception, breast-feeding, or patients who test positive for pregnancy at enrollment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2010-07; Primary Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Assessing safety through toxicities observed using CTCAE version 3.0 | At each study visit for the duration of the 12-week cycle

SECONDARY OUTCOMES:
Evaluating lesions using Response Evaluation Criteria in Solid Tumors (RECIST 1.0) | Every 8 weeks after treatment
Immunological responses to the treatment measured through analysis of blood draws | At the end of the 12-week cycle

CONTACTS AND LOCATIONS:
Overall Officials: Srikala Sridhar, MD FRCPC, Principal Investigator — University Health Network - Princess Margaret Hospital
Locations (1):
- Princess Margaret Hospital, Toronto, Ontario, Canada